CLINICAL TRIAL: NCT05058703
Title: Saraiki Translation, Validity & Reliability of the Activities Specific Balance Confidence (ABC) Scale Questionnaire in Older Adults
Brief Title: Saraiki Translation, Validity & Reliability of the Activities Specific Balance Confidence (ABC) Scale Questionnaire
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC01038 Farva Ikram
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Old Age; Debility
Keywords: balance; older adults
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a need for a culturally adapted screening tool to aid health care professionals or clinicians screen for the presence of fall and balance issues associated with injuries in saraiki population. Furthermore, while culturally adapting the scale is necessary, it is important that changes do not alter the original intent, which requires it to be broad, comprehensible and applicable to the entire population. As saraiki language is the most-used language in the South Punjab, translating and adapting the ABC scale to the saraiki population while accounting for its sociocultural characteristics is an important task. So, I decided to conduct a tool translation and validation study. This study will help the clinicians to assess their patient's confidence and balance easily through the saraiki version of ABC scale in saraiki population and hence will help in timely management of the balance.

DETAILED DESCRIPTION:
The ABC scale is a 16-item questionnaire with 11-point subscales that assess the level of confidence in performing a specific task without losing balance or becoming unsteady. Each item score ranges from 0% (no confidence) to 100% (total confidence).

As cross-border and cross-cultural studies continue to increase, there is a greater need for linguistic validation of tools across a variety of societies. Until now, no translation or adaptation of the ABC scale has been made for the population with different languages in Pakistan. In order to use questionnaires in areas with different languages and cultures, translation into new languages of ABC scale, for identifying fall and balance issues is required.

ELIGIBILITY:
Inclusion Criteria:

* Able to read saraiki language.
* Healthy older population
* People with controlled Diabetes mellitus
* People with controlled hypertension
* Older adults with BBS score 45-56.

Exclusion Criteria:

* Unstable medical condition.
* Cognitive issues like not able to concentrate, can't perform the task attentively.
* Any physical disability like not able to walk and patient with vestibular disorders.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older Adults
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Saraiki version of Activities-specific Balance Confidence Scale | 1 week
  The ABC scale is a 16-item questionnaire with 11-point subscales that assess the level of confidence in performing a specific task without losing balance or becoming unsteady. Each item score ranges from 0% (no confidence) to 100% (total confidence) and the total score of the S-ABC is obtained by adding up the ratings (0-160) and then dividing by 16
Twelve Item Short Form Health Survey (SF-12) | 1 week
  The 12-item Short Form Health Survey (SF-12) is a multipurpose, generic, 12-item questionnaire developed from the Short Form Health Survey 36 (SF-36). The SF-12 generates a Physical Component Summary scale score (PCS-SF12) and a Mental Component Summary scale score (MCS-SF12). Several studies have reported its validity and reliability as a measure of health-related quality of life in different populations.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Civil Hospital, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No